CLINICAL TRIAL: NCT05609474
Title: Trajectories and Reactions of Users and Relatives Consulting French Youth Addiction Services (Consultations Jeunes Consommateurs)
Brief Title: Trajectories and Reactions of Users and Relatives Consulting French Youth Addiction Services
Acronym: TRYAD
Status: Recruiting | Type: Observational
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01365-36
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Addiction
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Users (adolescents or young adults): 1430 users (adolescents and young adults) with addiction problems and consulting CJC for the first time
- Caregivers: 715 caregivers
- Consultations Jeunes Consommateurs CJCs: Initial survey (month 0) of participating CJCs: assessment of the "structural" characteristics of the CJCs (type of CJC (hospital, association), urban/rural area, number of users, number of consultations per month, type of workers...)
  - Telephone interview at the 6th and 12th month: assessment of variables related to the user's pathway (referral to a specialized medical or social service…)

SUMMARY:
In France, the "Consultations Jeunes Consommateurs" (CJC) are the services specialized in the reception of young people for addiction problems. There are more than 500 CJCs throughout France. Depending on the situation, the CJC develops an early intervention strategy aimed either at reducing the risk of developing an addiction or at accelerating entry into appropriate care. The CJCs also meet with family members or professionals who may also independently request help or advice.

Set up by the State since 2004, the action of the CJCs has never been formally evaluated. Only descriptive studies, carried out by the French Observatory of Drugs and Drug Addiction (OFDT), have made it possible to better understand the profile of people who consult CJCs. However, no longitudinal study has yet been carried out to understand the factors associated with the overall evolution of users consulting CJCs, nor with the level of satisfaction of users and those around them. Such objectives are complex, due to the diversity of situations encountered in CJCs and the heterogeneity of the CJCs themselves.

DETAILED DESCRIPTION:
This multicenter study will be open to 19 CJC (Consultations jeunes Consommateurs), based on a pre-selection by the partners of structures that are particularly willing to participate in the study (Fédération Addictions, Addictions-France).

However, other CJCs may be included depending on the progress of recruitment.

This recruitment of additional CJCs will be stratified to target a sample of CJCs representative of the CJCs on the metropolitan territory on the following characteristics:

* Region (13 major regions)
* Rural or urban area, as defined by INSEE
* Number of annual consultations

ELIGIBILITY:
Inclusion Criteria:

For users :

* First consultation in CJC
* From 12 to 25 years old

For caregivers :

* First consultation in CJC (with or without the youth) or second consultation if accompanying a user
* ≥ 18 ans

Exclusion Criteria:

* inability to reach by phone
* Insufficient french level

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Young people with addiction problems
Sampling Method: Probability Sample
Enrollment: 1430 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Evolution in Global Appraisal of Individual Needs Short Screener (GAIN-SS) score from first assessment to 12-month assessment | Two days ( at month 0 and month 12)
  The GAIN-SS scale is a self-administered questionnaire whose responses will be collected by telephone in a standardized manner for all included participants

SECONDARY OUTCOMES:
For users: Measurement of satisfaction with CJC use, assessed at 12 months, using the Client Satisfaction Questionnaire - 8 (CSQ-8) | One day (at month 12)
  Evaluation of the secondary criterion: Client Satisfaction Questionnaire - 8 (CSQ-8)
For caregivers : Measurement of satisfaction with CJC use, assessed at 12 months, using the Client Satisfaction Questionnaire - 8 (CSQ-8) | One day (at month 12)
  Client Satisfaction Questionnaire - 8 (CSQ-8)
For caregivers : Evolution in Strengths and Difficulties Questionnaire (SDQ) score from first assessment to 12-month assessment | Two days (at month 0 and month 12)
  Strengths and Difficulties Questionnaire (SDQ)
For all subjects included : Qualitative study : to assess their experience of the CJC's contribution to their needs and expectations | One day (month 12)
  Qualitative study on a sub-sample of caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin ROLLAND, PhD, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, Auvergne-Rhône-Alpes, France